CLINICAL TRIAL: NCT07300644
Title: A Randomized, Double-blind, Positive-controlled Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of 24-valent Pneumococcal Conjugate Vaccine in Children Aged 2 Months (Minimum 42 Days) to 5 Years
Brief Title: Clinical Trial of PCV24 in Infants and Children Aged 2 Months to 5 Years
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PCV24-1005
Record Dates: First submitted 2025-11-24; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pneumococcal Infectious Disease
Keywords: PCV24; Phase 2
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinovac PCV24 (Experimental): Sinovac PCV24 (0.5 mL) is administered intramuscularly according to different immunization schedules.
  Interventions: Biological: Sinovac PCV24
- Prevnar® (Active Comparator): Prevnar® (0.5 mL) is administered intramuscularly according to different immunization schedules.
  Interventions: Biological: Prevnar®

INTERVENTIONS:
Biological: Sinovac PCV24 — Sinovac PCV24 (0.5 mL) is administered intramuscularly according to different immunization schedules.
  Arms: Sinovac PCV24
Biological: Prevnar® — Prevnar® (0.5 mL) is administered intramuscularly according to different immunization schedules.
  Arms: Prevnar®

SUMMARY:
A Phase 2 clinical trial of 24-valent pneumococcal conjugate vaccine (PCV24) developed by Sinovac Life Science Co., Ltd will be conducted in the pediatric population aged 2 months (minimum 42 days) to 5 years.

The objective of the study is to evaluate the safety and immunogenicity of Sinovac PCV24. The trial is a randomized, double-blind, positive controlled phase 2 clinical trial.

DETAILED DESCRIPTION:
A phase 2 clinical trial of the study of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV24) developed by Sinovac Life Science Co., Ltd (Sinovac) will be conducted in the Chinese pediatric population aged 2 months (minimum 42 days) to 5 years. The trial is a randomized, double-blind, positive-controlled study. The objective of this study is to evaluate the safety and immunogenicity of PCV24 manufactured by Sinovac Life Science Co., Ltd. The active control vaccine is Prevenar13®, manufactured by Pfizer.

A total of at least 420 participants aged 2 months (minimum 42 days) to 5 years will be enrolled. Participants will be randomized in a 1:1 ratio to the test group and control group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants who are aged 2 months (42-89 days), 7-11 months, 12-23 months, and 2-5 years;
2. The participants' guardian provides a legal identity document and the participants' vaccination record;
3. The participant's guardian understands and voluntarily signs the informed consent form;
4. Follow all study procedures and stay in contact during the study.

Exclusion Criteria:

1. Received any pneumococcal vaccine prior to enrollment;
2. History of invasive pneumococcal diseases or other pneumococcal diseases caused by Streptococcus pneumoniae, as confirmed by laboratory tests;
3. History of severe adverse reactions to the vaccine or vaccine components, or history of allergy, such as urticaria, dyspnea, angioneurotic edema, anaphylactic shock;
4. Low birth weight (<2.5kg), or premature infant (gestation weeks < 37 weeks) (applies to infants younger than 12 months);
5. History of abnormal labor during delivery (planned cesarean section is excluded), history of asphyxia rescue and nervous system damage (applies to infants younger than 12 months);
6. Severe congenital malformations or developmental disorders, genetic defects, or malnutrition;
7. Have uncontrolled chronic diseases or history of severe diseases, including but not limited to cardiovascular diseases (e.g. congenital heart disease), hematological diseases (e.g. severe anemia), liver and kidney diseases, digestive diseases, respiratory diseases (such as active tuberculosis), malignant tumors and major functional organ transplantation history;
8. Autoimmune diseases, immunodeficiency diseases (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, autoimmune thyroid disease, asplenia, functional asplenia, HIV infection);
9. Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelet levels);
10. Have/have suffered from a serious neurological disorder (epilepsy or convulsions, but a febrile convulsion is not an exclusion criteria ) or mental illness, or have a family history of such diseases;
11. Consecutively received immunosuppressive therapy (excluding corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-concurrent dermatitis), or other immunoregulatory therapies, or cytotoxic therapy over 14 days within 6 months before vaccination, or plans to receive such therapies during the study;
12. Receipt of immunoglobulins or other blood products within 3 months prior to administration of the investigational vaccine (except for hepatitis B immunoglobulin or rabies immunoglobulin used within 1 month), or planned use of such products during the study period;
13. Received other investigational drugs or vaccines within 30 days prior to enrollment, or plan to receive such drugs or vaccines during the study;
14. Received live attenuated vaccine within 14 days prior to enrollment;
15. Received subunit or inactivated vaccine within 7 days prior to enrollment;
16. Acute diseases or acute onset of chronic diseases within 7 days prior to enrollment, known or potentially active infection;
17. Axillary temperature≥ 37.3 Degree Celsius before vaccination;
18. In the investigator's judgment, the participant has any other factors that make him or her unfit to participate in the clinical trial.

Ages: 42 Days to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) | 30 days after primary vaccination
Incidence of adverse reactions | 0-30 days after vaccination

SECONDARY OUTCOMES:
Pneumococcal serotype-specific IgG antibody geometric mean increase (GMI) | 30 days after the 2nd dose of the primary vaccination (2-month-olds), 30 days after primary vaccination (all participants)
OPA antibody levels for each pneumococcal serotype | 30 days after vaccination
Incidence of adverse reactions | 0-7 days after vaccination
Incidence of serious adverse events (SAE) | from vaccination to 6 months after final dose

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Qichun District Center for Disease Prevention and Control, Huanggang, Hubei
  - Xiangzhou District Center for Disease Prevention and Control, Xiangyang, Hubei
  - Xian'an District Center for Disease Prevention and Control, Xianning, Hubei

IPD SHARING:
Plan to Share IPD: No